CLINICAL TRIAL: NCT00862966
Title: Randomized Control Trial on Citrate as the Central Venous Catheter Lock Solution
Brief Title: Central Venous Catheter Lock Solution
Acronym: CVCLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center, Tuzla (Other)
Responsible Party: UNIVERSITY MEDICAL CENTER, Department of Dialysis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UMC-02-139
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia | interventions — Citric Acid; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- citrate (Experimental)
  Interventions: Other: citrate
- heparin (Active Comparator)
  Interventions: Other: heparin

INTERVENTIONS:
Other: citrate — comparison of different catheter lock solutions
  Arms: citrate
Other: heparin — comparison of different lock solutions
  Arms: heparin

SUMMARY:
The purpose of this study is to determine whether the application of 47% citrate lock solution decreases the incidence of infection and thrombosis of central venous catheter in hemodialysis population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of end stage renal disease

Exclusion Criteria:

* Patients refusing randomization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
lower incidence of infection | 1 year

SECONDARY OUTCOMES:
lower incidence of thrombosis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dialysis, Tuzla, TK, Bosnia and Herzegovina